CLINICAL TRIAL: NCT06566976
Title: Prehabilitation and Rehabilitation in PAD: A Randomized Exercise Intervention Trial (PREPARE-IT)
Brief Title: Prehabilitation and Rehabilitation in PAD
Acronym: PREPARE-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jonathan Myers, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYE0018APR
Record Dates: First submitted 2024-08-13; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prehabilitation (Experimental): Subjects randomized to the prehabilitation group will undergo 6 weeks of individualized exercise therapy, including a 1-week ramp-up period (3 sessions) conducted at the VAPAHCS rehabilitation facility. Subjects will then exercise primarily at home, with an in-clinic exercise session repeated weekly for the duration of their participation. These sessions will be individualized based on tolerance and in accordance with standardized guidelines, but will generally consist of 45-60 min of supervised exercise that combines aerobic and resistance training, including warm-up and cool-down. Throughout the study, subjects will be asked to perform 30 minutes of daily unsupervised aerobic exercise of their choice, with an emphasis on improving walking performance at home. Guidelines for patient monitoring, safety, and prescription outlined by the American Heart Association, American College Sports Medicine, and American Association of Cardiovascular and Pulmonary Rehabilitation will be followed.
  Interventions: Other: Exercise Intervention; Other: VAPAHCS Rehabilitation Core Components
- Rehabilitation (Active Comparator): Subjects randomized to the rehabilitation group will initiate exercise sessions approximately 2-weeks following endovascular intervention as outlined in guidelines for PAD. Patient stability and wound patency will be paramount considerations prior to a patient beginning the rehabilitation program. Similar to prehabilitation, subjects will undergo a 1-week, 3 session familiarization period conducted at the VAPAHCS rehabilitation facility, then return once weekly for in-clinic supervised sessions. The weekly in-person visits will be conducted at the rehabilitation center to monitor and encourage compliance, review activity questionnaires, download accelerometry data, and address any clinical concerns. Similar to participants in the prehabilitation group, the 6-week rehabilitation period will be individualized and follow standardized guidelines designed for rehabilitation in patients with PAD.
  Interventions: Other: Exercise Intervention; Other: VAPAHCS Rehabilitation Core Components
- Prehabiliation and Rehabilitation (Experimental): Subjects randomized to the prehabilitation and rehabilitation group will undergo both the 6 weeks of prehabilitation pre-operative and 6 weeks of rehabilitation post-operative as described in their respective arm descriptions.
  Interventions: Other: Exercise Intervention; Other: VAPAHCS Rehabilitation Core Components

INTERVENTIONS:
Other: Exercise Intervention — Aerobic and resistance exercise will be components of the prehabiliation and rehabilitation programs. Given the presence of PAD, a particular emphasis will be placed on volume of walking and improving walking performance.
  Other Names: Exercise Therapy
Other: VAPAHCS Rehabilitation Core Components — The prehabilitation and rehabilitation programs include all Core Components of rehabilitation as outlined in guidelines. The current clinical VAPAHCS program includes smoking cessation, nutrition, risk factor management and psychosocial counseling referrals as appropriate, and these services will be available for the current proposal.

SUMMARY:
To determine the effectiveness of pre and post-operative exercise therapy in patients undergoing peripheral artery stenting for peripheral arterial disease.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a form of cardiovascular disease that affects the arteries supplying blood flow to the legs. The prevalence of PAD is increasing rapidly in the United States. When PAD is severe, it can cause pain with movement and limit a person's ability to walk or perform their normal daily activities. With severe PAD, a procedure is often performed in which an artery is held open with a small tube called a stent.

Programs of exercise-based rehabilitation have been shown to greatly help these patients in terms of the pain they experience with walking, their ability to perform daily activities or those required by work, and improved quality of life. There is also a newer form of therapy, called prehabilitation, which has been shown to have important benefits for patients with PAD. Prehabilitation involves four to six weeks of exercise therapy and lifestyle recommendations before undergoing a stent procedure. Prehabilitation helps patients improve exercise tolerance and make lifestyle changes that improve risk factors before the procedure. Those who participate in prehabilitation programs have fewer complications with the stent procedure, spend fewer days in the hospital, and have a better ability to exercise and return to work more quickly.

Although the benefits of prehabilitation and rehabilitation are well established, most doctors neglect to recommend these treatments to their patients who undergo a stent procedure for PAD. The research team will study the impact of prehabilitation, rehabilitation or both forms of therapy. The results will likely encourage more doctors to recommend the best option for their patients, and possibly to recommend both prehabilitation and rehabilitation among patients who are having a stent procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female adult diagnosed with peripheral artery disease (PAD)
* Experiencing leg pain while walking
* Scheduled to have a stent for PAD
* Able to perform exercise safely
* Postmenopausal and not of child bearing capacity

Exclusion Criteria:

* Medically unstable patients
* Recent MI within 3 months
* Malignancy
* Uncontrolled diabetes mellitus (HBA1C ≥8 mmol/l)
* Alcoholism or other recreational drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Time to claudication pain | Baseline, 6 weeks, 14 weeks, 22 weeks
  Time to initial onset of claudication pain with exercise treadmill test.

SECONDARY OUTCOMES:
Peak VO2 | Baseline, 6 weeks, 14 weeks, 22 weeks
  Peak V02 will be determined on a treadmill using an individualized ramp protocol with collection of continuous ventilatory gas exchange responses.
6-minute walk test (6MWT) | Baseline, 6 weeks, 14 weeks, 22 weeks
  Total distance (meters) of walk in 6 minutes.
Walking Impairment Questionnaire (WIQ) | Baseline, 6 weeks, 14 weeks, 22 weeks
  Developed to evaluate walking limitations in patients with PAD. Assesses the ability of individuals to walk defined distances and speeds and climb stairs.
Peripheral Artery Questionnaire (PAQ) | Baseline, 6 weeks, 14 weeks, 22 weeks
  20-item questionnaire developed and validated specifically for PAD and is designed to quantify patients' physical limitations, symptoms, social function, treatment satisfaction, and quality of life.
Walking | Up to 22 weeks
  Physical activity patterns, expressed as steps/day will be quantified using fitness/health tracking device.
Energy expenditure | Up to 22 weeks
  Energy expenditure will be quantified using fitness/health tracking device.
Chair raises | Baseline, 6 weeks, 14 weeks, 22 weeks
  Number of repetitions completed within 60 seconds (46cm high seat).
Upper body strength | Baseline, 6 weeks, 14 weeks, 22 weeks
  1 repetition max for Chest Press.
Lower body strength | Baseline, 6 weeks, 14 weeks, 22 weeks
  1 repetition max for Leg Extension.
Hand grip strength | Baseline, 6 weeks, 14 weeks, 22 weeks
  Maximum isometric strength will be measured using a hand grip dynamometer.
Insulin sensitivity | Baseline, 6 weeks, 14 weeks, 22 weeks
  Fasting glucose and insulin samples will be obtained from blood draw to generate Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) score.
Lipid panel | Baseline, 6 weeks, 14 weeks, 22 weeks
  Fasting total cholesterol, LDL, HDL and triglycerides will be assessed from blood draw.
Sodium | Baseline, 6 weeks, 14 weeks, 22 weeks
  Standard Chem 20 blood draw will be used to obtain sodium in blood value.
Homocysteine | Baseline, 6 weeks, 14 weeks, 22 weeks
  Homocysteine will be assessed from blood draw.
High-sensitivity C-reactive protein (hs-CRP) | Baseline, 6 weeks, 14 weeks, 22 weeks
  High-sensitivity C-reactive protein (hs-CRP) will be assessed from blood draw.
Interleukin-6 (IL-6) | Baseline, 6 weeks, 14 weeks, 22 weeks
  Interleukin-6 (IL-6) will be assessed from blood draw.
D-dimer | Baseline, 6 weeks, 14 weeks, 22 weeks
  D-dimer will be assessed from blood draw.
Blood protein | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain blood protein value.
Albumin | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain albumin in blood value.
Calcium | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain calcium in blood value.
Potassium | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain potassium in blood value.
Chloride | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain chloride in blood value.
Carbon dioxide | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain carbon dioxide in blood value.
AST/GOTU/l | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain AST/GOTU/l in blood value.
ALT/GPT | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain ALT/GPT in blood value.
ALK Phosphatase | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain ALT/GPT in blood value.
Bilirubin | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain total bilirubin in blood value.
Urea Nitrogen | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain urea nitrogen in blood value.
Creatinine | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain creatinine in blood value.
eGFR | Baseline, 6 weeks, 14 weeks, 22 weeks
  Blood draw will be used to obtain eGFR value.

OTHER OUTCOMES:
Endothelial function | Baseline, 6 weeks, 14 weeks, 22 weeks
  The Endo Pat 2000 system will be used to perform this procedure. Both forearms will be occluded with a standard blood pressure cuff for 5 minutes.
Ankle-brachial index (ABI) | Baseline, 6 weeks, 14 weeks, 22 weeks
  Using a standard brachial artery cuff method with a Doppler ultrasound probe at the posterior tibial artery to determine ABI.
Exercise Benefits and Barriers Scale (EBBS) | Baseline, 6 weeks, 14 weeks, 22 weeks
  Perceived barriers and benefits to physical activity will be assessed using two methods: a semi-structured interview and administration of the Exercise Benefits and Barriers Scale (EBBS), to obtain both open-ended qualitative and quantitative data on these constructs. The EBBS may be used in its entirety or as two seperate scales. As a whole, scoring for EBBS ranges from 43 to 172 with a higher score being the individual perceives exercise more positively. When the Benefits Scale is used alone, the score range is between 29 to 116 with the higher the score being the individual perceives exercise more positively. When the Barriers Scale is used alone, the score range is between 14 to 56. The higher the score on the Barriers Scale, the greater the perception of barriers to exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] Correction. Circ Res. 2015 Jun 19;117(1):e12. doi: 10.1161/RES.0000000000000059. No abstract available. PMID 26089368
- [Background] Mayfield JA, Reiber GE, Maynard C, Czerniecki J, Sangeorzan B. The epidemiology of lower-extremity disease in veterans with diabetes. Diabetes Care. 2004 May;27 Suppl 2:B39-44. doi: 10.2337/diacare.27.suppl_2.b39. PMID 15113781
- [Background] Shu J, Santulli G. Update on peripheral artery disease: Epidemiology and evidence-based facts. Atherosclerosis. 2018 Aug;275:379-381. doi: 10.1016/j.atherosclerosis.2018.05.033. Epub 2018 May 22. No abstract available. PMID 29843915
- [Background] Horvath L, Nemeth N, Feher G, Kives Z, Endrei D, Boncz I. Epidemiology of Peripheral Artery Disease: Narrative Review. Life (Basel). 2022 Jul 12;12(7):1041. doi: 10.3390/life12071041. PMID 35888129
- [Background] Garg PK, Liu K, Tian L, Guralnik JM, Ferrucci L, Criqui MH, Tan J, McDermott MM. Physical activity during daily life and functional decline in peripheral arterial disease. Circulation. 2009 Jan 20;119(2):251-60. doi: 10.1161/CIRCULATIONAHA.108.791491. Epub 2008 Dec 31. PMID 19118256
- [Background] McDermott MM, Greenland P, Liu K, Guralnik JM, Criqui MH, Dolan NC, Chan C, Celic L, Pearce WH, Schneider JR, Sharma L, Clark E, Gibson D, Martin GJ. Leg symptoms in peripheral arterial disease: associated clinical characteristics and functional impairment. JAMA. 2001 Oct 3;286(13):1599-606. doi: 10.1001/jama.286.13.1599. PMID 11585483
- [Background] McDermott MM, Liu K, Ferrucci L, Tian L, Guralnik JM, Liao Y, Criqui MH. Greater sedentary hours and slower walking speed outside the home predict faster declines in functioning and adverse calf muscle changes in peripheral arterial disease. J Am Coll Cardiol. 2011 Jun 7;57(23):2356-64. doi: 10.1016/j.jacc.2010.12.038. PMID 21636037
- [Background] Hamburg NM, Balady GJ. Exercise rehabilitation in peripheral artery disease: functional impact and mechanisms of benefits. Circulation. 2011 Jan 4;123(1):87-97. doi: 10.1161/CIRCULATIONAHA.109.881888. No abstract available. PMID 21200015
- [Background] Myers JN, Fonda H. The Impact of Fitness on Surgical Outcomes: The Case for Prehabilitation. Curr Sports Med Rep. 2016 Jul-Aug;15(4):282-9. doi: 10.1249/JSR.0000000000000274. PMID 27399826
- [Background] Myers J, Niebauer J, Humphrey R. Prehabilitation Coming of Age: IMPLICATIONS FOR CARDIAC AND PULMONARY REHABILITATION. J Cardiopulm Rehabil Prev. 2021 May 1;41(3):141-146. doi: 10.1097/HCR.0000000000000574. PMID 33512981
- [Background] Cheng XS, Myers JN, Chertow GM, Rabkin R, Chan KN, Chen Y, Tan JC. Prehabilitation for kidney transplant candidates: Is it time? Clin Transplant. 2017 Aug;31(8). doi: 10.1111/ctr.13020. Epub 2017 Jul 10. PMID 28564126
- [Background] Brunelli A, Kim AW, Berger KI, Addrizzo-Harris DJ. Physiologic evaluation of the patient with lung cancer being considered for resectional surgery: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e166S-e190S. doi: 10.1378/chest.12-2395. PMID 23649437
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 9;130(24):e278-333. doi: 10.1161/CIR.0000000000000106. Epub 2014 Aug 1. No abstract available. PMID 25085961
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, Gan TJ, Kennedy RH, Ljungqvist O, Lobo DN, Miller T, Radtke FF, Ruiz Garces T, Schricker T, Scott MJ, Thacker JK, Ytrebo LM, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice. Acta Anaesthesiol Scand. 2016 Mar;60(3):289-334. doi: 10.1111/aas.12651. Epub 2015 Oct 30. PMID 26514824
- [Background] Ljungqvist O, Francis N, Urman R (Eds.). Enhanced Recovery After Surgery. A Complete Guide to Optimizing Outcomes. New York: Springer, 2020.
- [Background] Orange ST, Northgraves MJ, Marshall P, Madden LA, Vince RV. Exercise prehabilitation in elective intra-cavity surgery: A role within the ERAS pathway? A narrative review. Int J Surg. 2018 Aug;56:328-333. doi: 10.1016/j.ijsu.2018.04.054. Epub 2018 May 3. PMID 29730070
- [Background] Thomas SG, Marzolini S, Lin E, Nguyen CH, Oh P. Peripheral Arterial Disease: Supervised Exercise Therapy Through Cardiac Rehabilitation. Clin Geriatr Med. 2019 Nov;35(4):527-537. doi: 10.1016/j.cger.2019.07.009. Epub 2019 Jul 2. PMID 31543183
- [Background] Devrome AN, Aggarwal S, McMurtry MS, Southern D, Hauer T, Lamb B, Arena R, Moore RD, Wilton SB, Stone J, Martin BJ. Cardiac rehabilitation in people with peripheral arterial disease: A higher risk population that benefits from completion. Int J Cardiol. 2019 Jun 15;285:108-114. doi: 10.1016/j.ijcard.2019.02.070. Epub 2019 Mar 5. PMID 30857844
- [Background] Stewart KJ, Hiatt WR, Regensteiner JG, Hirsch AT. Exercise training for claudication. N Engl J Med. 2002 Dec 12;347(24):1941-51. doi: 10.1056/NEJMra021135. No abstract available. PMID 12477945
- [Background] Murphy TP, Cutlip DE, Regensteiner JG, Mohler ER, Cohen DJ, Reynolds MR, Massaro JM, Lewis BA, Cerezo J, Oldenburg NC, Thum CC, Goldberg S, Jaff MR, Steffes MW, Comerota AJ, Ehrman J, Treat-Jacobson D, Walsh ME, Collins T, Badenhop DT, Bronas U, Hirsch AT; CLEVER Study Investigators. Supervised exercise versus primary stenting for claudication resulting from aortoiliac peripheral artery disease: six-month outcomes from the claudication: exercise versus endoluminal revascularization (CLEVER) study. Circulation. 2012 Jan 3;125(1):130-9. doi: 10.1161/CIRCULATIONAHA.111.075770. Epub 2011 Nov 16. PMID 22090168
- [Background] Spronk S, Bosch JL, den Hoed PT, Veen HF, Pattynama PM, Hunink MG. Intermittent claudication: clinical effectiveness of endovascular revascularization versus supervised hospital-based exercise training--randomized controlled trial. Radiology. 2009 Feb;250(2):586-95. doi: 10.1148/radiol.2501080607. PMID 19188327
- [Background] Kruidenier LM, Nicolai SP, Rouwet EV, Peters RJ, Prins MH, Teijink JA. Additional supervised exercise therapy after a percutaneous vascular intervention for peripheral arterial disease: a randomized clinical trial. J Vasc Interv Radiol. 2011 Jul;22(7):961-8. doi: 10.1016/j.jvir.2011.02.017. Epub 2011 May 14. PMID 21571547
- [Background] Olin JW, White CJ, Armstrong EJ, Kadian-Dodov D, Hiatt WR. Peripheral Artery Disease: Evolving Role of Exercise, Medical Therapy, and Endovascular Options. J Am Coll Cardiol. 2016 Mar 22;67(11):1338-57. doi: 10.1016/j.jacc.2015.12.049. PMID 26988957
- [Background] Olin JW, Sealove BA. Peripheral artery disease: current insight into the disease and its diagnosis and management. Mayo Clin Proc. 2010 Jul;85(7):678-92. doi: 10.4065/mcp.2010.0133. PMID 20592174
- [Background] McDermott MM, Guralnik JM, Ferrucci L, Tian L, Liu K, Liao Y, Green D, Sufit R, Hoff F, Nishida T, Sharma L, Pearce WH, Schneider JR, Criqui MH. Asymptomatic peripheral arterial disease is associated with more adverse lower extremity characteristics than intermittent claudication. Circulation. 2008 May 13;117(19):2484-91. doi: 10.1161/CIRCULATIONAHA.107.736108. Epub 2008 May 5. PMID 18458172
- [Background] Regensteiner JG, Hiatt WR, Coll JR, Criqui MH, Treat-Jacobson D, McDermott MM, Hirsch AT. The impact of peripheral arterial disease on health-related quality of life in the Peripheral Arterial Disease Awareness, Risk, and Treatment: New Resources for Survival (PARTNERS) Program. Vasc Med. 2008 Feb;13(1):15-24. doi: 10.1177/1358863X07084911. PMID 18372434
- [Background] Smolderen KG, Hoeks SE, Pedersen SS, van Domburg RT, de Liefde II, Poldermans D. Lower-leg symptoms in peripheral arterial disease are associated with anxiety, depression, and anhedonia. Vasc Med. 2009 Nov;14(4):297-304. doi: 10.1177/1358863X09104658. PMID 19808714
- [Background] Gardner AW, Montgomery PS, Parker DE. Physical activity is a predictor of all-cause mortality in patients with intermittent claudication. J Vasc Surg. 2008 Jan;47(1):117-22. doi: 10.1016/j.jvs.2007.09.033. PMID 18178462
- [Background] McDermott MM, Tian L, Liu K, Guralnik JM, Ferrucci L, Tan J, Pearce WH, Schneider JR, Criqui MH. Prognostic value of functional performance for mortality in patients with peripheral artery disease. J Am Coll Cardiol. 2008 Apr 15;51(15):1482-9. doi: 10.1016/j.jacc.2007.12.034. PMID 18402904
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Watson L, Ellis B, Leng GC. Exercise for intermittent claudication. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD000990. doi: 10.1002/14651858.CD000990.pub2. PMID 18843614
- [Background] van den Houten MM, Lauret GJ, Fakhry F, Fokkenrood HJ, van Asselt AD, Hunink MG, Teijink JA. Cost-effectiveness of supervised exercise therapy compared with endovascular revascularization for intermittent claudication. Br J Surg. 2016 Nov;103(12):1616-1625. doi: 10.1002/bjs.10247. Epub 2016 Aug 11. PMID 27513296
- [Background] Spronk S, Bosch JL, den Hoed PT, Veen HF, Pattynama PM, Hunink MG. Cost-effectiveness of endovascular revascularization compared to supervised hospital-based exercise training in patients with intermittent claudication: a randomized controlled trial. J Vasc Surg. 2008 Dec;48(6):1472-80. doi: 10.1016/j.jvs.2008.06.016. Epub 2008 Sep 4. PMID 18771879
- [Background] Reynolds MR, Apruzzese P, Galper BZ, Murphy TP, Hirsch AT, Cutlip DE, Mohler ER 3rd, Regensteiner JG, Cohen DJ. Cost-effectiveness of supervised exercise, stenting, and optimal medical care for claudication: results from the Claudication: Exercise Versus Endoluminal Revascularization (CLEVER) trial. J Am Heart Assoc. 2014 Nov 11;3(6):e001233. doi: 10.1161/JAHA.114.001233. PMID 25389284
- [Background] Mouch CA, Kenney BC, Lorch S, Montgomery JR, Gonzalez-Walker M, Bishop K, Palazzolo WC, Sullivan JA, Wang SC, Englesbe MJ. Statewide Prehabilitation Program and Episode Payment in Medicare Beneficiaries. J Am Coll Surg. 2020 Mar;230(3):306-313.e6. doi: 10.1016/j.jamcollsurg.2019.10.014. Epub 2019 Dec 5. PMID 31812662
- [Background] Santa Mina D, Scheede-Bergdahl C, Gillis C, Carli F. Optimization of surgical outcomes with prehabilitation. Appl Physiol Nutr Metab. 2015 Sep;40(9):966-9. doi: 10.1139/apnm-2015-0084. Epub 2015 May 13. PMID 26300015
- [Background] Jack S, West M, Grocott MP. Perioperative exercise training in elderly subjects. Best Pract Res Clin Anaesthesiol. 2011 Sep;25(3):461-72. doi: 10.1016/j.bpa.2011.07.003. PMID 21925410
- [Background] Levett DZ, Grocott MP. Cardiopulmonary exercise testing, prehabilitation, and Enhanced Recovery After Surgery (ERAS). Can J Anaesth. 2015 Feb;62(2):131-42. doi: 10.1007/s12630-014-0307-6. Epub 2015 Jan 22. PMID 25608638
- [Background] Barakat HM, Shahin Y, Barnes R, Gohil R, Souroullas P, Khan J, McCollum PT, Chetter IC. Supervised exercise program improves aerobic fitness in patients awaiting abdominal aortic aneurysm repair. Ann Vasc Surg. 2014 Jan;28(1):74-9. doi: 10.1016/j.avsg.2013.09.001. PMID 24332259
- [Background] Nagarajan K, Bennett A, Agostini P, Naidu B. Is preoperative physiotherapy/pulmonary rehabilitation beneficial in lung resection patients? Interact Cardiovasc Thorac Surg. 2011 Sep;13(3):300-2. doi: 10.1510/icvts.2010.264507. Epub 2011 May 17. PMID 21586476
- [Background] Myers JN, White JJ, Narasimhan B, Dalman RL. Effects of exercise training in patients with abdominal aortic aneurysm: preliminary results from a randomized trial. J Cardiopulm Rehabil Prev. 2010 Nov-Dec;30(6):374-83. doi: 10.1097/HCR.0b013e3181ebf2db. PMID 20724934
- [Background] Myers J, McElrath M, Jaffe A, Smith K, Fonda H, Vu A, Hill B, Dalman R. A randomized trial of exercise training in abdominal aortic aneurysm disease. Med Sci Sports Exerc. 2014 Jan;46(1):2-9. doi: 10.1249/MSS.0b013e3182a088b8. PMID 23793234
- [Background] Smith TB, Stonell C, Purkayastha S, Paraskevas P. Cardiopulmonary exercise testing as a risk assessment method in non cardio-pulmonary surgery: a systematic review. Anaesthesia. 2009 Aug;64(8):883-93. doi: 10.1111/j.1365-2044.2009.05983.x. PMID 19604193
- [Background] Smith JL, Verrill TA, Boura JA, Sakwa MP, Shannon FL, Franklin BA. Effect of cardiorespiratory fitness on short-term morbidity and mortality after coronary artery bypass grafting. Am J Cardiol. 2013 Oct 15;112(8):1104-9. doi: 10.1016/j.amjcard.2013.05.057. Epub 2013 Jul 10. PMID 23849973
- [Background] Shaarani SR, Moyna N, Moran R, O'Byrne JM. Prehabilitation: The void in the management of anterior cruciate ligament injuries-A Clinical Review. ISRN Rehabilitation. 2012;1-11:938974.
- [Background] O'Doherty AF, West M, Jack S, Grocott MP. Preoperative aerobic exercise training in elective intra-cavity surgery: a systematic review. Br J Anaesth. 2013 May;110(5):679-89. doi: 10.1093/bja/aes514. Epub 2013 Feb 7. PMID 23393151
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Mar 21;69(11):1465-1508. doi: 10.1016/j.jacc.2016.11.008. Epub 2016 Nov 13. No abstract available. PMID 27851991
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Firnhaber JM, Powell CS. Lower Extremity Peripheral Artery Disease: Diagnosis and Treatment. Am Fam Physician. 2019 Mar 15;99(6):362-369. PMID 30874413
- [Background] Shammas NW. Epidemiology, classification, and modifiable risk factors of peripheral arterial disease. Vasc Health Risk Manag. 2007;3(2):229-34. doi: 10.2147/vhrm.2007.3.2.229. PMID 17580733
- [Background] Biccard BM, Nepaul S. Risk factors associated with intermediate and long-term mortality following vascular surgery in South African patients. Cardiovasc J Afr. 2010 Sep-Oct;21(5):263-7. doi: 10.5830/cvja-2010-016. PMID 20972514
- [Background] Bertges DJ, Goodney PP, Zhao Y, Schanzer A, Nolan BW, Likosky DS, Eldrup-Jorgensen J, Cronenwett JL; Vascular Study Group of New England. The Vascular Study Group of New England Cardiac Risk Index (VSG-CRI) predicts cardiac complications more accurately than the Revised Cardiac Risk Index in vascular surgery patients. J Vasc Surg. 2010 Sep;52(3):674-83, 683.e1-683.e3. doi: 10.1016/j.jvs.2010.03.031. Epub 2010 Jun 8. PMID 20570467
- [Background] Banta MR, Ma F, Bravata DM, Kirsner RS, Federman DG. Incidence of and factors associated with achieving target lipid levels in patients with peripheral arterial disease. J Gen Intern Med. 2006 Jul;21(7):711-4. doi: 10.1111/j.1525-1497.2006.00456.x. PMID 16808771
- [Background] Vouri SM, Shaw RF, Waterbury NV, Egge JA, Alexander B. Prevalence of achievement of A1c, blood pressure, and cholesterol (ABC) goal in veterans with diabetes. J Manag Care Pharm. 2011 May;17(4):304-12. doi: 10.18553/jmcp.2011.17.4.304. PMID 21534641
- [Background] Sandesara PB, Lambert CT, Gordon NF, Fletcher GF, Franklin BA, Wenger NK, Sperling L. Cardiac rehabilitation and risk reduction: time to "rebrand and reinvigorate". J Am Coll Cardiol. 2015 Feb 3;65(4):389-395. doi: 10.1016/j.jacc.2014.10.059. PMID 25634839
- [Background] Balady GJ, Williams MA, Ades PA, Bittner V, Comoss P, Foody JM, Franklin B, Sanderson B, Southard D; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Epidemiology and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism; American Association of Cardiovascular and Pulmonary Rehabilitation. Core components of cardiac rehabilitation/secondary prevention programs: 2007 update: a scientific statement from the American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; the Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; and the American Association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2007 May 22;115(20):2675-82. doi: 10.1161/CIRCULATIONAHA.106.180945. Epub 2007 May 18. PMID 17513578
- [Background] McCullough PA, Gallagher MJ, Dejong AT, Sandberg KR, Trivax JE, Alexander D, Kasturi G, Jafri SM, Krause KR, Chengelis DL, Moy J, Franklin BA. Cardiorespiratory fitness and short-term complications after bariatric surgery. Chest. 2006 Aug;130(2):517-25. doi: 10.1378/chest.130.2.517. PMID 16899853
- [Background] Powers SK, Quindry JC, Kavazis AN. Exercise-induced cardioprotection against myocardial ischemia-reperfusion injury. Free Radic Biol Med. 2008 Jan 15;44(2):193-201. doi: 10.1016/j.freeradbiomed.2007.02.006. Epub 2007 Feb 21. PMID 18191755
- [Background] Pitsavos C, Kavouras SA, Panagiotakos DB, Arapi S, Anastasiou CA, Zombolos S, Stravopodis P, Mantas Y, Kogias Y, Antonoulas A, Stefanadis C; GREECS Study Investigators. Physical activity status and acute coronary syndromes survival The GREECS (Greek Study of Acute Coronary Syndromes) study. J Am Coll Cardiol. 2008 May 27;51(21):2034-9. doi: 10.1016/j.jacc.2008.01.053. PMID 18498957
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Background] Nielsen PR, Jorgensen LD, Dahl B, Pedersen T, Tonnesen H. Prehabilitation and early rehabilitation after spinal surgery: randomized clinical trial. Clin Rehabil. 2010 Feb;24(2):137-48. doi: 10.1177/0269215509347432. PMID 20103575
- [Background] Tung-Chou Li, Ming-Chung Yang, Ailun Heather Tseng, Henry Hsin-Chung Lee, Prehabilitation and rehabilitation for surgically treated lung cancer patients, Journal of Cancer Research and Practice. 2017;4:89-94.
- [Background] Parashar S, Spertus JA, Tang F, Bishop KL, Vaccarino V, Jackson CF, Boyden TF, Sperling L. Predictors of early and late enrollment in cardiac rehabilitation, among those referred, after acute myocardial infarction. Circulation. 2012 Sep 25;126(13):1587-95. doi: 10.1161/CIRCULATIONAHA.111.088799. Epub 2012 Aug 28. PMID 22929302
- [Background] Brady S, Purdham D, Oh P, Grace S. Clinical and sociodemographic correlates of referral for cardiac rehabilitation following cardiac revascularization in Ontario. Heart Lung. 2013 Sep-Oct;42(5):320-5. doi: 10.1016/j.hrtlng.2013.07.001. PMID 23998380
- [Background] Chang P, Nead KT, Olin JW, Myers J, Cooke JP, Leeper NJ. Effect of physical activity assessment on prognostication for peripheral artery disease and mortality. Mayo Clin Proc. 2015 Mar;90(3):339-45. doi: 10.1016/j.mayocp.2014.12.016. Epub 2015 Jan 31. PMID 25649965
- [Background] Brown R. Review of Article: Leeper, N.J., Myers, J., Zhou, M., Nead, K.T., Syed, A., Kojima, Y. ... Cooke, J.P. (2013). Exercise capacity is the strongest predictor of mortality in patients with peripheral arterial disease. Journal of Vascular Surgery, 57, 728-33. J Vasc Nurs. 2017 Jun;35(2):112-113. doi: 10.1016/j.jvn.2017.04.002. Epub 2017 Apr 28. No abstract available. PMID 28527724
- [Background] Hankey GJ, Norman PE, Eikelboom JW. Medical treatment of peripheral arterial disease. JAMA. 2006 Feb 1;295(5):547-53. doi: 10.1001/jama.295.5.547. PMID 16449620
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Hiatt WR, Fowkes FG, Heizer G, Berger JS, Baumgartner I, Held P, Katona BG, Mahaffey KW, Norgren L, Jones WS, Blomster J, Millegard M, Reist C, Patel MR; EUCLID Trial Steering Committee and Investigators. Ticagrelor versus Clopidogrel in Symptomatic Peripheral Artery Disease. N Engl J Med. 2017 Jan 5;376(1):32-40. doi: 10.1056/NEJMoa1611688. Epub 2016 Nov 13. PMID 27959717
- [Background] Gardner AW, Katzel LI, Sorkin JD, Bradham DD, Hochberg MC, Flinn WR, Goldberg AP. Exercise rehabilitation improves functional outcomes and peripheral circulation in patients with intermittent claudication: a randomized controlled trial. J Am Geriatr Soc. 2001 Jun;49(6):755-62. doi: 10.1046/j.1532-5415.2001.49152.x. PMID 11454114
- [Background] Spronk S, Bosch JL, Veen HF, den Hoed PT, Hunink MG. Intermittent claudication: functional capacity and quality of life after exercise training or percutaneous transluminal angioplasty--systematic review. Radiology. 2005 Jun;235(3):833-42. doi: 10.1148/radiol.2353040457. Epub 2005 Apr 28. PMID 15860674
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): executive summary a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease) endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. J Am Coll Cardiol. 2006 Mar 21;47(6):1239-312. doi: 10.1016/j.jacc.2005.10.009. No abstract available. PMID 16545667
- [Background] Lourenco ALG, da Silva JL, Leite JC. The impact of peripheral arterial disease on exercise tolerance and quality of life in the elderly and the role of cardiovascular physiotherapy: review article. J Vasc Bras. 2021 Apr 28;20:e20200117. doi: 10.1590/1677-5449.200117. PMID 34093682
- [Background] Myers, J. Essentials of Cardiopulmonary Exercise Testing. Champaign: Human Kinetics, 1996.
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Kanakaraj M, Yates DR, Wilson RJT, Baroni ML, Davies SJ. Prognostic Markers of Outcome in Patients Undergoing Infra-inguinal Revascularisation: A Prospective Observational Pilot Study. Eur J Vasc Endovasc Surg. 2017 Aug;54(2):212-219. doi: 10.1016/j.ejvs.2017.05.005. Epub 2017 Jun 16. PMID 28625356
- [Background] Montgomery PS, Gardner AW. The clinical utility of a six-minute walk test in peripheral arterial occlusive disease patients. J Am Geriatr Soc. 1998 Jun;46(6):706-11. doi: 10.1111/j.1532-5415.1998.tb03804.x. PMID 9625185
- [Background] McDermott MM, Guralnik JM, Criqui MH, Liu K, Kibbe MR, Ferrucci L. Six-minute walk is a better outcome measure than treadmill walking tests in therapeutic trials of patients with peripheral artery disease. Circulation. 2014 Jul 1;130(1):61-8. doi: 10.1161/CIRCULATIONAHA.114.007002. No abstract available. PMID 24982117
- [Background] Nayak P, Guralnik JM, Polonsky TS, Kibbe MR, Tian L, Zhao L, Criqui MH, Ferrucci L, Li L, Zhang D, McDermott MM. Association of six-minute walk distance with subsequent lower extremity events in peripheral artery disease. Vasc Med. 2020 Aug;25(4):319-327. doi: 10.1177/1358863X20901599. Epub 2020 Apr 27. PMID 32338582
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] American Association of Cardiovascular and Pulmonary Rehabilitation. Guidelines for Cardiac Rehabilitation and Secondary Prevention Programs, (5th ed). Champaign: Human Kinetics, 2020.
- [Background] Stewart K, Franklin B, Squires R. Resistance training in patients with CHD. In Graves JE and Franklin BA, Resistance Training in Health and Rehabilitation. Champaign: Human Kinetics, pp217-236,2001.
- [Background] Thurston B, Dawson J. Ankle Brachial Pressure Index: An update for the vascular specialist and general practitioner. Vascular. 2019 Oct;27(5):560-570. doi: 10.1177/1708538119842395. Epub 2019 Apr 5. No abstract available. PMID 30952202
- [Background] Brevetti G, Silvestro A, Di Giacomo S, Bucur R, Di Donato A, Schiano V, Scopacasa F. Endothelial dysfunction in peripheral arterial disease is related to increase in plasma markers of inflammation and severity of peripheral circulatory impairment but not to classic risk factors and atherosclerotic burden. J Vasc Surg. 2003 Aug;38(2):374-9. doi: 10.1016/s0741-5214(03)00124-1. PMID 12891123
- [Background] Pande RL, Perlstein TS, Beckman JA, Creager MA. Association of insulin resistance and inflammation with peripheral arterial disease: the National Health and Nutrition Examination Survey, 1999 to 2004. Circulation. 2008 Jul 1;118(1):33-41. doi: 10.1161/CIRCULATIONAHA.107.721878. Epub 2008 Jun 16. PMID 18559705
- [Background] Hirsch AT, Gotto AM Jr. Undertreatment of dyslipidemia in peripheral arterial disease and other high-risk populations: an opportunity for cardiovascular disease reduction. Vasc Med. 2002;7(4):323-31. doi: 10.1191/1358863x02vm453ra. PMID 12710848
- [Background] Tzoulaki I, Murray GD, Lee AJ, Rumley A, Lowe GD, Fowkes FG. C-reactive protein, interleukin-6, and soluble adhesion molecules as predictors of progressive peripheral atherosclerosis in the general population: Edinburgh Artery Study. Circulation. 2005 Aug 16;112(7):976-83. doi: 10.1161/CIRCULATIONAHA.104.513085. Epub 2005 Aug 8. PMID 16087797
- [Background] Saetre T, Enoksen E, Lyberg T, Stranden E, Jorgensen JJ, Sundhagen JO, Hisdal J. Supervised exercise training reduces plasma levels of the endothelial inflammatory markers E-selectin and ICAM-I in patients with peripheral arterial disease. Angiology. 2011 May;62(4):301-5. doi: 10.1177/0003319710385338. PMID 21474466
- [Background] McDermott MM, Liu K, Ferrucci L, Tian L, Guralnik JM, Green D, Tan J, Liao Y, Pearce WH, Schneider JR, McCue K, Ridker P, Rifai N, Criqui MH. Circulating blood markers and functional impairment in peripheral arterial disease. J Am Geriatr Soc. 2008 Aug;56(8):1504-10. doi: 10.1111/j.1532-5415.2008.01797.x. Epub 2008 Jul 24. PMID 18662216
- [Background] Woo KS, Chook P, Lolin YI, Cheung AS, Chan LT, Sun YY, Sanderson JE, Metreweli C, Celermajer DS. Hyperhomocyst(e)inemia is a risk factor for arterial endothelial dysfunction in humans. Circulation. 1997 Oct 21;96(8):2542-4. doi: 10.1161/01.cir.96.8.2542. PMID 9355891
- [Background] Abdellaoui A, Al-Khaffaf H. C-reactive protein (CRP) as a marker in peripheral vascular disease. Eur J Vasc Endovasc Surg. 2007 Jul;34(1):18-22. doi: 10.1016/j.ejvs.2006.10.040. Epub 2007 Feb 12. PMID 17296319
- [Background] Collins TC, Lunos S, Carlson T, Henderson K, Lightbourne M, Nelson B, Hodges JS. Effects of a home-based walking intervention on mobility and quality of life in people with diabetes and peripheral arterial disease: a randomized controlled trial. Diabetes Care. 2011 Oct;34(10):2174-9. doi: 10.2337/dc10-2399. Epub 2011 Aug 26. PMID 21873560
- [Background] McDermott MM, Ades P, Guralnik JM, Dyer A, Ferrucci L, Liu K, Nelson M, Lloyd-Jones D, Van Horn L, Garside D, Kibbe M, Domanchuk K, Stein JH, Liao Y, Tao H, Green D, Pearce WH, Schneider JR, McPherson D, Laing ST, McCarthy WJ, Shroff A, Criqui MH. Treadmill exercise and resistance training in patients with peripheral arterial disease with and without intermittent claudication: a randomized controlled trial. JAMA. 2009 Jan 14;301(2):165-74. doi: 10.1001/jama.2008.962. PMID 19141764
- [Background] Nicolai SP, Kruidenier LM, Rouwet EV, Graffius K, Prins MH, Teijink JA. The walking impairment questionnaire: an effective tool to assess the effect of treatment in patients with intermittent claudication. J Vasc Surg. 2009 Jul;50(1):89-94. doi: 10.1016/j.jvs.2008.12.073. PMID 19563956
- [Background] Sagar SP, Brown PM, Zelt DT, Pickett WL, Tranmer JE. Further clinical validation of the walking impairment questionnaire for classification of walking performance in patients with peripheral artery disease. Int J Vasc Med. 2012;2012:190641. doi: 10.1155/2012/190641. Epub 2012 Aug 2. PMID 22919494
- [Background] Nead KT, Zhou M, Diaz Caceres R, Olin JW, Cooke JP, Leeper NJ. Walking impairment questionnaire improves mortality risk prediction models in a high-risk cohort independent of peripheral arterial disease status. Circ Cardiovasc Qual Outcomes. 2013 May 1;6(3):255-61. doi: 10.1161/CIRCOUTCOMES.111.000070. Epub 2013 Apr 30. PMID 23633217
- [Background] Spertus J, Jones P, Poler S, Rocha-Singh K. The peripheral artery questionnaire: a new disease-specific health status measure for patients with peripheral arterial disease. Am Heart J. 2004 Feb;147(2):301-8. doi: 10.1016/j.ahj.2003.08.001. PMID 14760329
- [Background] McDermott MM, Greenland P, Guralnik JM, Liu K, Criqui MH, Pearce WH, Chan C, Schneider J, Sharma L, Taylor LM, Arseven A, Quann M, Celic L. Depressive symptoms and lower extremity functioning in men and women with peripheral arterial disease. J Gen Intern Med. 2003 Jun;18(6):461-7. doi: 10.1046/j.1525-1497.2003.20527.x. PMID 12823653
- [Background] Arya S, Lee S, Zahner GJ, Cohen BE, Hiramoto J, Wolkowitz OM, Khakharia A, Binney ZO, Grenon SM. The association of comorbid depression with mortality and amputation in veterans with peripheral artery disease. J Vasc Surg. 2018 Aug;68(2):536-545.e2. doi: 10.1016/j.jvs.2017.10.092. Epub 2018 Mar 24. PMID 29588133
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Ramirez JL, Grenon SM. Depression and peripheral artery disease: why we should care and what we can do. CVIR Endovasc. 2018;1(1):14. doi: 10.1186/s42155-018-0017-1. Epub 2018 Sep 18. No abstract available. PMID 30652146
- [Background] Sechrist KR, Walker SN, Pender NJ. Development and psychometric evaluation of the exercise benefits/barriers scale. Res Nurs Health. 1987 Dec;10(6):357-65. doi: 10.1002/nur.4770100603. PMID 3423307
- [Background] Whipple MO, Schorr EN, Talley KMC, Lindquist R, Bronas UG, Treat-Jacobson D. A mixed methods study of perceived barriers to physical activity, geriatric syndromes, and physical activity levels among older adults with peripheral artery disease and diabetes. J Vasc Nurs. 2019 Jun;37(2):91-105. doi: 10.1016/j.jvn.2019.02.001. Epub 2019 Mar 11. PMID 31155168
- [Background] Myers J, Kaykha A, George S, Abella J, Zaheer N, Lear S, Yamazaki T, Froelicher V. Fitness versus physical activity patterns in predicting mortality in men. Am J Med. 2004 Dec 15;117(12):912-8. doi: 10.1016/j.amjmed.2004.06.047. PMID 15629729
- [Background] Myers J, Dupain M, Vu A, Jaffe A, Smith K, Fonda H, Dalman R. Agreement between activity-monitoring devices during home rehabilitation: a substudy of the AAA STOP trial. J Aging Phys Act. 2014 Jan;22(1):87-95. doi: 10.1123/japa.2012-0133. Epub 2013 Feb 14. PMID 23416349
- [Background] Myers J, Chan K, Chen Y, Lit Y, Patti A, Massaband P, Kiratli BJ, Tamura M, Chertow GM, Rabkin R. Effect of a Home-Based Exercise Program on Indices of Physical Function and Quality of Life in Elderly Maintenance Hemodialysis Patients. Kidney Blood Press Res. 2021;46(2):196-206. doi: 10.1159/000514269. Epub 2021 Mar 26. PMID 33774634
- [Background] ACSM Guidelines for Exercise Testing and Exercise Prescription, 9th edition. Baltimore: LW&W, 2021.
- [Background] Myers J. Principles of exercise prescription for patients with chronic heart failure. Heart Fail Rev. 2008 Feb;13(1):61-8. doi: 10.1007/s10741-007-9051-0. PMID 17939037
- [Background] Borg GAV. Borg's Perceived Exertion and Pain Scales. Champaign, IL: Human Kinetics, 1998.
- [Background] Christopherson DJ, Phillips WT, Louie D. Effect of resistance training with Therabands on function ability and strength in cardiac rehabilitation participants. J Cardiopulm Rehabil. 1998;5:372-376.
- [Background] Ata R, Gandhi N, Rasmussen H, El-Gabalawy O, Gutierrez S, Ahmad A, Suresh S, Ravi R, Rothenberg K, Aalami O. Clinical validation of smartphone-based activity tracking in peripheral artery disease patients. NPJ Digit Med. 2018 Dec 11;1:66. doi: 10.1038/s41746-018-0073-x. eCollection 2018. PMID 31304343
- [Background] Liang G, Huang X, Hirsch J, Mehmi S, Fonda H, Chan K, Huang NF, Aalami O, Froelicher VF, Lee DP, Myers J, Lee AS, Nguyen PK. Modest Gains After an 8-Week Exercise Program Correlate With Reductions in Non-traditional Markers of Cardiovascular Risk. Front Cardiovasc Med. 2021 Jun 17;8:669110. doi: 10.3389/fcvm.2021.669110. eCollection 2021. PMID 34222367
- [Background] Arena R, Myers J, Williams MA, Gulati M, Kligfield P, Balady GJ, Collins E, Fletcher G; American Heart Association Committee on Exercise, Rehabilitation, and Prevention of the Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Nursing. Assessment of functional capacity in clinical and research settings: a scientific statement from the American Heart Association Committee on Exercise, Rehabilitation, and Prevention of the Council on Clinical Cardiology and the Council on Cardiovascular Nursing. Circulation. 2007 Jul 17;116(3):329-43. doi: 10.1161/CIRCULATIONAHA.106.184461. Epub 2007 Jun 18. No abstract available. PMID 17576872
- [Background] Myers J, Buchanan N, Walsh D, Kraemer M, McAuley P, Hamilton-Wessler M, Froelicher VF. Comparison of the ramp versus standard exercise protocols. J Am Coll Cardiol. 1991 May;17(6):1334-42. doi: 10.1016/s0735-1097(10)80144-5. PMID 2016451
- [Background] Froelicher V, Myers J. Exercise and the Heart. St Louis, WB Saunders, pp. 249-250, 2006.
- [Background] Shue P, Froelicher V. EXTRA: An expert system for exercise test reporting. J Non-Invas Test. 1998;II-4: 21-27.
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Background] Lane R, Harwood A, Watson L, Leng GC. Exercise for intermittent claudication. Cochrane Database Syst Rev. 2017 Dec 26;12(12):CD000990. doi: 10.1002/14651858.CD000990.pub4. PMID 29278423
- [Background] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997
- [Background] Gardner AW, Montgomery PS, Wang M. Minimal clinically important differences in treadmill, 6-minute walk, and patient-based outcomes following supervised and home-based exercise in peripheral artery disease. Vasc Med. 2018 Aug;23(4):349-357. doi: 10.1177/1358863X18762599. Epub 2018 Apr 19. PMID 29671381
- [Background] McElrath M, Myers J, Chan K, Fonda H. Exercise adherence in the elderly: Experience with abdominal aortic aneurysm simple treatment and prevention. J Vasc Nurs. 2017 Mar;35(1):12-20. doi: 10.1016/j.jvn.2016.08.002. PMID 28224946
- [Background] Hallgren KA, Witkiewitz K. Missing data in alcohol clinical trials: a comparison of methods. Alcohol Clin Exp Res. 2013 Dec;37(12):2152-60. doi: 10.1111/acer.12205. Epub 2013 Jul 24. PMID 23889334
- [Background] Witkiewitz K, Falk DE, Kranzler HR, Litten RZ, Hallgren KA, O'Malley SS, Anton RF; Alcohol Clinical Trials Initiative (ACTIVE) Workgroup. Methods to analyze treatment effects in the presence of missing data for a continuous heavy drinking outcome measure when participants drop out from treatment in alcohol clinical trials. Alcohol Clin Exp Res. 2014 Nov;38(11):2826-34. doi: 10.1111/acer.12543. PMID 25421518
- [Background] Jackson D, White IR, Mason D, Sutton S. A general method for handling missing binary outcome data in randomized controlled trials. Addiction. 2014 Dec;109(12):1986-93. doi: 10.1111/add.12721. PMID 25171441
- [Background] Myers J, Ahnve S, Froelicher V, Livingston M, Jensen D, Abramson I, Sullivan M, Mortara D. A randomized trail of the effects of 1 year of exercise training on computer-measured ST segment displacement in patients with coronary artery disease. J Am Coll Cardiol. 1984 Dec;4(6):1094-102. doi: 10.1016/s0735-1097(84)80127-8. PMID 6389645
- [Background] Myers J, Gademan M, Brunner K, Kottman W, Boesch C, Dubach P. Effects of high-intensity training on indices of ventilatory efficiency in chronic heart failure. J Cardiopulm Rehabil Prev. 2012 Jan-Feb;32(1):9-16. doi: 10.1097/HCR.0b013e3182343bdf. PMID 22113369
- [Background] Myers J, Wagner D, Schertler T, Beer M, Luchinger R, Klein M, Rickli H, Muller P, Mayer K, Schwitter J, Dubach P. Effects of exercise training on left ventricular volumes and function in patients with nonischemic cardiomyopathy: application of magnetic resonance myocardial tagging. Am Heart J. 2002 Oct;144(4):719-25. doi: 10.1067/mhj.2002.124401. PMID 12360170
- [Background] Dunlay SM, Witt BJ, Allison TG, Hayes SN, Weston SA, Koepsell E, Roger VL. Barriers to participation in cardiac rehabilitation. Am Heart J. 2009 Nov;158(5):852-9. doi: 10.1016/j.ahj.2009.08.010. Epub 2009 Sep 29. PMID 19853708
- [Background] Sun V, Raz DJ, Kim JY, Melstrom L, Hite S, Varatkar G, Fong Y. Barriers and facilitators of adherence to a perioperative physical activity intervention for older adults with cancer and their family caregivers. J Geriatr Oncol. 2020 Mar;11(2):256-262. doi: 10.1016/j.jgo.2019.06.003. Epub 2019 Jun 14. PMID 31208829
- [Background] Birtwistle SB, Jones I, Murphy R, Gee I, Watson PM. Family support for physical activity post-myocardial infarction: A qualitative study exploring the perceptions of cardiac rehabilitation practitioners. Nurs Health Sci. 2021 Mar;23(1):227-236. doi: 10.1111/nhs.12806. Epub 2021 Jan 26. PMID 33389812
- [Background] Arena R, Williams M, Forman DE, Cahalin LP, Coke L, Myers J, Hamm L, Kris-Etherton P, Humphrey R, Bittner V, Lavie CJ; American Heart Association Exercise, Cardiac Rehabilitation and Prevention Committee of the Council on Clinical Cardiology, Council on Epidemiology and Prevention, and Council on Nutrition, Physical Activity and Metabolism. Increasing referral and participation rates to outpatient cardiac rehabilitation: the valuable role of healthcare professionals in the inpatient and home health settings: a science advisory from the American Heart Association. Circulation. 2012 Mar 13;125(10):1321-9. doi: 10.1161/CIR.0b013e318246b1e5. Epub 2012 Jan 30. No abstract available. PMID 22291128
- [Background] Treat-Jacobson D, McDermott MM, Bronas UG, Campia U, Collins TC, Criqui MH, Gardner AW, Hiatt WR, Regensteiner JG, Rich K; American Heart Association Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Council on Cardiovascular and Stroke Nursing. Optimal Exercise Programs for Patients With Peripheral Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Jan 22;139(4):e10-e33. doi: 10.1161/CIR.0000000000000623. No abstract available. PMID 30586765
- [Background] American Association of Cardiovascular and Pulmonary Rehabilitation; American College of Cardiology Foundation; American Heart Association Task Force on Performance Measures (Writing Committee to Develop Clinical Performance Measures for Cardiac Rehabilitation); Thomas RJ, King M, Lui K, Oldridge N, Pina IL, Spertus J. AACVPR/ACCF/AHA 2010 Update: Performance Measures on Cardiac Rehabilitation for Referral to Cardiac Rehabilitation/Secondary Prevention Services Endorsed by the American College of Chest Physicians, the American College of Sports Medicine, the American Physical Therapy Association, the Canadian Association of Cardiac Rehabilitation, the Clinical Exercise Physiology Association, the European Association for Cardiovascular Prevention and Rehabilitation, the Inter-American Heart Foundation, the National Association of Clinical Nurse Specialists, the Preventive Cardiovascular Nurses Association, and the Society of Thoracic Surgeons. J Am Coll Cardiol. 2010 Sep 28;56(14):1159-67. doi: 10.1016/j.jacc.2010.06.006. No abstract available. PMID 20863958
- [Background] Dubach P, Myers J, Dziekan G, Goebbels U, Reinhart W, Vogt P, Ratti R, Muller P, Miettunen R, Buser P. Effect of exercise training on myocardial remodeling in patients with reduced left ventricular function after myocardial infarction: application of magnetic resonance imaging. Circulation. 1997 Apr 15;95(8):2060-7. doi: 10.1161/01.cir.95.8.2060. PMID 9133516
- [Background] Dubach P, Myers J, Dziekan G, Goebbels U, Reinhart W, Muller P, Buser P, Stulz P, Vogt P, Ratti R. Effect of high intensity exercise training on central hemodynamic responses to exercise in men with reduced left ventricular function. J Am Coll Cardiol. 1997 Jun;29(7):1591-8. doi: 10.1016/s0735-1097(97)82540-5. PMID 9180124
- [Background] Myers J, Fonda H, Vasanawala M, Chung K, Segall G, Chan K, Nguyen P. PCI Alternative Using Sustained Exercise (PAUSE): Rationale and trial design. Contemp Clin Trials. 2019 Apr;79:37-43. doi: 10.1016/j.cct.2019.02.010. Epub 2019 Feb 20. PMID 30797041
- [Background] Campbell EB, Delgadillo M, Lazzeroni LC, Louras PN, Myers J, Yesavage J, Fairchild JK. Cognitive Improvement Following Physical Exercise and Cognitive Training Intervention for Older Adults With MCI. J Gerontol A Biol Sci Med Sci. 2023 Mar 1;78(3):554-560. doi: 10.1093/gerona/glac189. PMID 36099058
- [Background] Moore CS, Myers J, Yesavage JA, Fairchild JK. Ventilatory efficiency is associated with memory decay in older adults with amnestic mild cognitive impairment. Submitted, 2022
- [Background] Moore CS, Myers J, Yesavage JA, Fairchild JK. Assessment of physical activity in older adults with cognitive impairment. Submitted, 2022
- [Background] Fairchild JK, Myers J, Louras P, Jo B, McNerney MW, Salehi A, Hallmayer J, Yesavage J. A Combined physical and cognitive training program for veterans with mild cognitive impairment: A randomized clinical trial. Submitted, 2022.
- See also: U.S. Markets for Peripheral Vascular Stents — http://www.medtechinsight.com/ReportA254.html
- See also: Related Info — https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?NCAId=287
- See also: Wilson C, Colombo R. Association of Community Cancer Centers. Making the business case for implementing prehabilitation services — https://www.accc-cancer.org/docs/documents/meetings/ufo/ufo-2019-prehab-services-tool.pdf
- See also: Bloom E. Prehabilitation evidence and insight review. Macmillan National Cancer Rehabilitation, 2018. — https://www.macmillan.org.uk/_images/prehabilitation-evidence-and-insight-review_tcm9-335025.pdf
- See also: Centers for Medicare & Medicaid Services. Decision Memo for Supervised Exercise Therapy (SET) for Symptomatic Peripheral Artery Disease — https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?NCAId=287
- See also: Related Info — https://www.thesagegroup.us/reports/the-real-cost-of-peripheral-artery-disease/
- See also: Related Info — https://www.cms.gov/newsroom/fact-sheets/physician-quality-reporting-system-and-e-prescribing-program